CLINICAL TRIAL: NCT01004991
Title: Phase I/II Trial of Azacytidine + R-CHOP in Diffuse Large B-Cell Lymphoma
Brief Title: Phase I/II Trial of R-CHOP + Azacytidine in Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0907010513
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisone; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): subjects will receive azacytidine dose dependent on dose-escalation schedule at time of enrollment - all will receive standard dose RCHOP
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: vincristine; Drug: doxorubicin; Drug: prednisone; Drug: azacytidine

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 on Day 8 of each of 6 cycles
Drug: cyclophosphamide — 750 mg/m2 on Day 8 of each of 6 cycles
Drug: vincristine — 1.4 mg/m2 on Day 8 of each of 6 cycles
Drug: doxorubicin — 50 mg/m2 on Day 8 of each of 6 cycles
Drug: prednisone — 100 mg PO days 8-12 of each of 6 cycles
Drug: azacytidine — Dose level 1: azacytidine 25 mg/m2 days 1-5 Dose level 2: azacytidine 50 mg/m2 days 1-5 Dose level 3: azacytidine 75 mg/m2 days 1-5

SUMMARY:
This is a phase I/II open label, multi-center study of azacytidine in combination with standard RCHOP therapy in patients with DLBCL. Patients will be treated with azacytidine at escalating doses on days 1-5, followed by standard dose rituximab plus CHOP chemotherapy on day 8, every 21 days. Patients will be treated for a total 6 cycles. The phase II portion will then evaluate efficacy of the combination at the established MTD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed DLBCL with characteristic immunophenotypic profiles. Tumor tissue must be confirmed to express the CD20 antigen by flow cytometry or immunohistochemistry.
* Patients must have at least one site of measurable disease, 1.5 cm in diameter or greater.
* Patient has not had any previous treatment.
* Stage II (not appropriate for abbreviated chemoimmunotherapy and radiotherapy), III or IV disease
* Able to adhere to the study visit schedule and other protocol requirements.
* Patients must have laboratory test results within these ranges:

  * Absolute neutrophil count > = 1500/mm³
  * Platelet count > = 75,000/mm³
  * Serum creatinine < = 1.5X upper limit of normal (ULN)
  * Total bilirubin < = 1.5X ULN. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
  * AST (SGOT) and ALT (SGPT) < = 2 x ULN
* Disease free of prior malignancies for > = 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment.
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with azacitidine. The effects of azacytidine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Age >18 years.
* Ability to understand and the willingness to sign a written informed consent document.
* ECOG performance status of 0-2

Exclusion Criteria:

* Patients must not have any serious medical condition, laboratory abnormality,or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patients must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis B.
* Known central nervous system involvement by lymphoma.
* Known or suspected hypersensitivity to azacitidine or mannitol.
* Patients must not have advanced malignant hepatic tumors.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Complete Response
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 12
Participants | 11

ADVERSE EVENTS:
Groups:
- All Patients: all study patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=12)
Neutropenia (Blood and lymphatic system disorders) | 12
Neutropenic Fever (Blood and lymphatic system disorders) | 4
thrombocytopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes